CLINICAL TRIAL: NCT00818428
Title: The Contribution of a Speech Perception Intervention to the Prevention of Phonological Awareness Deficits in Children With Speech Sound Disorders
Brief Title: Randomized Clinical Trial of Phonological Interventions
Acronym: ECRIP
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: McGill University (Other)
Responsible Party: Susan Rvachew, Ph.D., S-LP(C), Associate Professor, Acting Director, School of Communication Sciences and Disorders, Faculty of Medicine, McGill University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: 410-2008-0503
Record Dates: First submitted 2009-01-05; First posted 2009-01-07 (Estimated); Last update posted 2009-09-23 (Estimated); Status verified 2009-09

CONDITIONS: Speech Articulation Disorder; Developmental Articulation Disorder; Phonological Impairment; Dyslexia
Keywords: Phonological Awareness; Speech Articulation Disorder; Development Articulation Disorder; Phonological Impairment; Dyslexia; Speech Therapy; School Transition
MeSH Terms: conditions — Articulation Disorders; Dyslexia; Communication Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Active Comparator): Speech Production Intervention + Articulation Parent Group
  Interventions: Behavioral: Speech Production Intervention; Behavioral: Articulation Parent Group
- 2 (Experimental): Speech Production Intervention + Dialogic Reading Parent Group
  Interventions: Behavioral: Speech Production Intervention; Behavioral: Dialogic Reading Parent Group
- 3 (Experimental): Speech Perception Intervention + Articulation Parent Group
  Interventions: Behavioral: Speech Perception Intervention; Behavioral: Articulation Parent Group
- 4 (Experimental): Speech Perception Intervention + Dialogical Reading Parent Group
  Interventions: Behavioral: Speech Perception Intervention; Behavioral: Dialogic Reading Parent Group

INTERVENTIONS:
Behavioral: Speech Production Intervention — Individual speech therapy directed at teaching the child to articulation specific speech sounds or word shapes accurately using traditional procedures such as phonetic placement and imitated and spontaneous speech production practice with feedback from the clinician about accuracy of articulatory gestures and knowledge of results.
  Other Names: Articulation therapy
  Arms: 1; 2
Behavioral: Speech Perception Intervention — Individualized intervention in which the Speech Assessment and Interactive Learning System is used to teach the child to identify recordings of words as either correct or incorrect pronunciations of the target word. In the event that the child is completely unable to pronounce the target speech sounds or word shapes focused stimulation activities are used to provide the child with further auditory exposure to the target forms. If the child stimulable for the target forms, the child is given opportunities the produce the target speech sounds or word shapes in the context of minimal pair games in which the child receives feedback about the communicative effectiveness of his or her attempts to produce the target words.
  Arms: 3; 4
Behavioral: Articulation Parent Group — Parents are taught to carry out home practice activities that focus on the child's ability to correctly articulate target speech sounds and word shapes.
  Arms: 1; 3
Behavioral: Dialogic Reading Parent Group — Parents are taught to read to their children using interactive techniques that help their children acquire new vocabulary, verbal reasoning abilities, and preliteracy skills.
  Arms: 2; 4

SUMMARY:
Recent research reveals genetic and symptomatic overlap among children with speech sound disorders (i.e., those who (misarticulate more sounds than would be expected for their age) and children with dyslexia (i.e., those who struggle to learn to read). Children who have speech sound disorders as preschoolers are at risk for the later emergence of dyslexia, a risk that often reveals itself in the form of poor phonological awareness skills during the preschool period. Traditional speech therapy methods focus on articulation accuracy and do not focus on the child's more abstract knowledge of the sound system of the language. The ultimate objective of this research program is to prevent reading disability in children who present with speech sounds disorders. The relative effectiveness of different interventions to help these children achieve age-appropriate phonological processing skills prior to school entry will be investigated. It is expected that a combination of treatment approaches that focus on speech perception skills and vocabulary knowledge will have a superior impact on phonological awareness in comparison with a treatment approach that focuses solely on articulation accuracy.

DETAILED DESCRIPTION:
The 72 children participating in the study will be randomly assigned (with concealment of the randomization sequence from study staff) to one of two Child Speech Interventions: Speech Perception or Speech Production. These interventions will be provided in individualized one-hour treatment sessions once per week for six consecutive weeks during the first treatment block. During the second 6 week treatment block all children will receive a group phonological awareness intervention. Concurrently their parents will be randomly assigned to receive instruction in the provision of a home program, either Articulation Therapy or Dialogic Reading. This will result in 4 groups of 18 children with each group receiving one of four combinations of intervention: Speech Production Intervention + Articulation Parent Group; Speech Production Intervention + Dialogic Reading Parent Group; Speech Perception Intervention + Articulation Parent Group; and Speech Perception Intervention + Dialogic Reading Parent Group. Assessments will occur pretreatment, after the first treatment block, after the second treatment block, and 9 months after the end of the second treatment block.

ELIGIBILITY:
Inclusion Criteria:

* primary diagnosis of speech articulation disorder/phonological impairment
* age 4 to 5 years of age at onset of treatment
* maternal language Canadian French (at least 75% exposure)
* must misarticulate at least two phonemes that would typically be mastered by their normally developing age peers

Exclusion Criteria:

* speech disorder is secondary to a primary condition (e.g., hearing impairment, cleft palate, autism, Down syndrome etc.)

Ages: 48 Months to 71 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 96 (Estimated)
Dates: Start 2008-11; Primary Completion 2010-07 (Estimated); Study Completion 2010-07 (Estimated)

PRIMARY OUTCOMES:
Phonological Awareness (Test d'Analyse Auditive en Français [Auditory Analysis Test in French]) | 12 months post treatment onset

SECONDARY OUTCOMES:
Articulation Accuracy (Test Francophone de Phonologie, Paul et Rvachew [Test of French Phonology) | 6 weeks post treatment onset; 12 weeks post-treatment onset; 12 months post-treatment onset
Vocabulary Knowledge (Échelle de Vocabulaire en Image Peabody [Peabody Picture Vocabulary Test - French Edition) | 12 months post-treatment onset
Phonological Awareness (Test de Conscience Phonologique, Brosseau-Lapre et Rvachew [Phonological Awareness Test - French Version]) | 6 weeks post-treatment onset; 12 weeks post-treatment onset

CONTACTS AND LOCATIONS:
Overall Officials: Susan Rvachew, Ph.D., Principal Investigator — McGill University
Locations (2):
- Canada (2):
  - McGill University, Montreal, Quebec
  - Montreal Children's Hospital, Montreal, Quebec